CLINICAL TRIAL: NCT05563766
Title: A Phase II Trial to Evaluate the Effect of Itraconazole on Pathologic Complete Response Rates in Resectable Esophageal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Durham VA Health Care System (U.S. Federal Agency); VA Palo Alto Health Care System (U.S. Federal Agency); Portland VA Medical Center (U.S. Federal Agency); VA Puget Sound Health Care System (U.S. Federal Agency); Michael E. DeBakey VA Medical Center (U.S. Federal Agency); VA Boston Healthcare System (U.S. Federal Agency); North Texas Veterans Healthcare System (U.S. Federal Agency); VA Ann Arbor Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONCB-016-21F; I01CX002349 (NIH)
Record Dates: First submitted 2022-09-27; First posted 2022-10-03 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Esophageal Adenocarcinoma; Esophageal Squamous Cell Carcinoma; Gastroesophageal Junction Carcinoma
Keywords: Itraconazole; Neoadjuvant
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — Itraconazole

STUDY DESIGN:
Intervention Model Description: Single arm, patients will receive itraconazole 300 mg po bid for two weeks prior and 6-8 weeks after standard of care neoadjuvant chemoradiation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Itraconazole (Experimental): Itraconazole 300 mg po bid for two weeks prior and 6-8 weeks after completion of standard of care neoadjuvant chemoradiation
  Interventions: Drug: Itraconazole

INTERVENTIONS:
Drug: Itraconazole — Itraconazole 300 mg po bid for two weeks prior and 6-8 weeks after completion of standard of care neoadjuvant chemoradiation

SUMMARY:
Esophageal cancer, which has a low 5-year overall survival rate (<20%) is increasing in incidence. Previous studies have shown that Hedgehog, AKT, and angiogenic signaling pathways are activated in a significant number of esophageal cancers. Itraconazole, a widely used anti-fungal medication, effectively inhibits these pathways. In this multi-site phase II trial, the investigators will evaluate the effect of itraconazole as a neoadjuvant therapy added to standard of care chemoradiation and surgery in the the treatment of locoregional esophageal and gastroesophageal junction cancers.

DETAILED DESCRIPTION:
Esophageal cancer has a high incidence rate in the United States, and novel approaches to improve its treatment are being studied. Itraconazole, an antifungal agent approved by the FDA in 1992, has been shown to inhibit the Hedgehog (Hh), AKT, and VEGFR2 signaling pathways which are upregulated in esophageal cancer and promote tumor growth. This study will evaluate whether the use of itraconazole leads to increased rates of pathologic complete response (pathCR) by at least 15% compared to propensity-score matched control patients with esophageal or gastroesophageal junction (GEJ) cancer. The investigators will enroll 78 patients with esophageal or GEJ cancer who will undergo standard of care staging workup with a PET/CT and endoscopic ultrasound (EUS). If no distant metastases are found, patients will receive 2 weeks of oral itraconazole before starting standard of care neoadjuvant chemoradiation. Upon completion of chemoradiation, patients will receive oral itraconazole for 6-8 weeks. Adverse effects to itraconazole will be monitored and drug levels will be obtained during clinic visits. If standard restaging PET/CT following neoadjuvant chemoradiation does not reveal new metastases, patients will undergo esophagectomy after consultation with their physician team. Samples from normal esophageal tissue will be analyzed for presence of itraconazole and its metabolite to determine if patients were compliant in taking study drug. Residual tumor tissue will be evaluated for status of the Hh, AKT, and VEGFR2 pathways with comparisons made to pre-treatment biopsies. The final pathology report will indicate whether the patient has achieved pathCR. Because Hh, AKT, and angiogenic signaling pathways can be upregulated in response to chemoradiation, the investigators believe that administering itraconazole around chemoradiation will lead to higher pathCR rates. This in turn should be able to improve treatment outcomes in patients with esophageal and GEJ cancer. Secondary endpoints include correlating drug levels and molecular pathway status to pathCR, determining a genomic profile that predicts treatment response, and evaluating ctDNA and exosomes as additional markers of treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving informed consent
* Pathologic diagnosis of esophageal cancer (ESCC or EAC) or GEJ cancer deemed resectable by a surgeon with a plan to undergo neoadjuvant chemoradiation and curative intent esophagectomy
* World Health Organization (WHO)/ECOG performance status (PS) of 0-2 at enrollment
* Adequate renal and liver function as judged by the treating physician

Exclusion Criteria:

* Inability to provide Informed Consent
* NYHA class III or IV CHF
* LFT>3X upper limit of normal
* Drug allergy to itraconazole
* Positive pregnancy test
* Those with QTc>450 ms will have QTc monitored during therapy by serial EKG to ensure QTc does not lengthen to what the treating clinician considers significant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-06-15 (Estimated)

PRIMARY OUTCOMES:
Rate of pathological complete response with itraconazole | 20 weeks
  Historically, the pathCR rate at time of esophagectomy is 25%. The investigators have powered our study to detect a 15% or more improvement in pathCR rate following treatment with itraconazole. By inhibiting pathways that mediate chemoradiation resistance, the investigators anticipate an improved pathCR rate.

SECONDARY OUTCOMES:
Comparison of Hedgehog, AKT, and angiogenesis pathway status before and after intervention | 20 weeks
  After completion of pathologic staging of any residual tumor at esophagectomy, FFPE sections will be analyzed for expression of SHH, GLI, HER2, phospho-S6, and CD34 by IHC or ISH and compared to untreated biopsies.
Correlation of peripheral blood and esophageal tissue levels of itraconazole and hydroxyitraconazole with pathologic response | 20 weeks
  Peripheral blood will be obtained during a standard of care clinic visit and squamous esophageal tissue collected at esophagectomy. These levels will be correlated with pathologic response.
Develop a predictive genomic profile of treatment response | 20 weeks
  Whole exome sequencing will be obtained on pre-treatment tumors from all enrolled patients. VA Boston HCS will use multiple algorithms to develop a genomic profile that predicts treatment response.
Determine the utility of ctDNA and exosome characterization as a prognostic marker | 20 weeks
  CtDNA will be obtained at 4 timepoints and exosomes will be collected at 3 timepoints during treatment. Changes in ctDNA quantitation and exosome characteristics will be correlated with pathologic treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: David H Wang, MD PhD, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (7):
- United States (7):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang W, Bhagwath AS, Ramzan Z, Williams TA, Subramaniyan I, Edpuganti V, Kallem RR, Dunbar KB, Ding P, Gong K, Geurkink SA, Beg MS, Kim J, Zhang Q, Habib AA, Choi SH, Lapsiwala R, Bhagwath G, Dowell JE, Melton SD, Jie C, Putnam WC, Pham TH, Wang DH. Itraconazole Exerts Its Antitumor Effect in Esophageal Cancer By Suppressing the HER2/AKT Signaling Pathway. Mol Cancer Ther. 2021 Oct;20(10):1904-1915. doi: 10.1158/1535-7163.MCT-20-0638. Epub 2021 Aug 10. PMID 34376577
- [Background] Kim J, Tang JY, Gong R, Kim J, Lee JJ, Clemons KV, Chong CR, Chang KS, Fereshteh M, Gardner D, Reya T, Liu JO, Epstein EH, Stevens DA, Beachy PA. Itraconazole, a commonly used antifungal that inhibits Hedgehog pathway activity and cancer growth. Cancer Cell. 2010 Apr 13;17(4):388-99. doi: 10.1016/j.ccr.2010.02.027. PMID 20385363
- [Background] Chen MB, Liu YY, Xing ZY, Zhang ZQ, Jiang Q, Lu PH, Cao C. Itraconazole-Induced Inhibition on Human Esophageal Cancer Cell Growth Requires AMPK Activation. Mol Cancer Ther. 2018 Jun;17(6):1229-1239. doi: 10.1158/1535-7163.MCT-17-1094. Epub 2018 Mar 28. PMID 29592879
- [Background] Kelly RJ, Ansari AM, Miyashita T, Zahurak M, Lay F, Ahmed AK, Born LJ, Pezhouh MK, Salimian KJ, Ng C, Matsangos AE, Stricker-Krongrad AH, Mukaisho KI, Marti GP, Chung CH, Canto MI, Rudek MA, Meltzer SJ, Harmon JW. Targeting the Hedgehog Pathway Using Itraconazole to Prevent Progression of Barrett's Esophagus to Invasive Esophageal Adenocarcinoma. Ann Surg. 2021 Jun 1;273(6):e206-e213. doi: 10.1097/SLA.0000000000003455. PMID 31290765